CLINICAL TRIAL: NCT01126151
Title: Parent Interventions to Prevent Student Drinking
Acronym: ACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Robert Turrisi, Professor, Penn State University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: R01AA015737 (NIH)
Record Dates: First submitted 2010-05-17; First posted 2010-05-19 (Estimated); Last update posted 2017-12-15 (Actual); Status verified 2017-12

CONDITIONS: Alcohol Consumption
Keywords: drinking; alcohol consequences
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- parent handbook (Experimental): parent handbook to increase the quantity and quality of communications about alcohol
  Interventions: Behavioral: parent handbook
- parent handbook with boosters (Experimental): boosters are given to parents at three times (move in, visit weekend; student visits home)
  Interventions: Behavioral: parent handbook
- parent handbook delay (Experimental): parent handbook is delayed and given after semester has begun
  Interventions: Behavioral: parent handbook

INTERVENTIONS:
Behavioral: parent handbook — parent handbook
  Other Names: Parent Communication Materials

SUMMARY:
Examine the efficacy of parent interventions to prevent college student drinking in first year students.

DETAILED DESCRIPTION:
The aims of the study are to:

1. efficacy of parent interventions to prevent college student drinking in first year students;
2. examine mediators of efficacy; and
3. examine moderators of efficacy.

ELIGIBILITY:
Inclusion Criteria:

* first year students

Exclusion Criteria:

* none

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1900 (Actual)
Dates: Start 2006-07; Primary Completion 2010-10 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
heavy episodic drinking | 12 months post baseline
  frequency of heavy episodic events

SECONDARY OUTCOMES:
drinking related consequences | 12 months post baseline
  Assess blackouts, hangovers, vomiting, fights, unplanned sex, academic problems and trouble with the police using the RAPI; YAAPST (standard assessment instruments for college alcohol prevention trials)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Turrisi, Ph.D., Principal Investigator — Penn State University
Locations (1):
- Penn State University, University Park, Pennsylvania, United States